CLINICAL TRIAL: NCT01266668
Title: Matched Pair Analysis Comparing the Outcomes of Primary Breast and Nodal Diffuse Large B Cell Lymphoma in Patients Treated With R-CHOP; Consortium for Improving Survival of Lymphoma (CISL) Study
Brief Title: The Impact of Rituximab in Patients With Primary Breast Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Ho-Young Yhim, Clinical professor, Chonbuk National University Hospital
Other Study IDs: Chonbuk 011
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Diffuse large B cell lymphoma; Breast; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary breast DLBCL: Primary breast DLBCL was defined as that involving single extranodal organ (i.e. breast) regardless of the status of nodal disease.
- Nodal DLBCL: The disease was only limited to the lymph nodes or lymphoid organs without extranodal organ involvements.

SUMMARY:
The purpose of this study is to investigate the impact of rituximab in primary breast DLBCL using a matched pair analysis following strict matching criteria in patients with primary breast and nodal DLBCL treated with rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) regimen.

DETAILED DESCRIPTION:
Primary breast lymphoma represents 1.7% to 2.2% of all extranodal non-Hodgkin's lymphoma. Histologically, the diffuse large B cell lymphoma (DLBCL) is the most predominant subtype of PBL. Previous studies in the pre-rituximab era have identified the worse outcomes in primary breast DLBCL compared with nodal DLBCL. Few clinical studies have been reported for investigating the efficacy of rituximab in patients with primary breast DLBCL. For clarifying this, a large randomized trial comparing survival in patients with primary breast DLBCL is required. However, the rarity of primary breast DLBCL makes large trial virtually difficult in single center or study group. Additionally, retrospective studies for evaluating the role of rituximab in primary breast DLBCL had bias according to the difference of treatment period between CHOP and R-CHOP era. Thus, in attempt to clarify the impact of rituximab on survival and patterns of progression in patients with primary breast DLBCL, the investigators performed this matched pair analysis following strict matching criteria in patients with primary breast DLBCL, who were identified from our previous nation-wide survey, and nodal DLBCL, who were selected from the data registry of Korean Society of Hematology Lymphoma Working Party, treated with R-CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Stage I or II of primary breast DLBCL treated with R-CHOP
* Stage I or II of nodal DLBCL treated with R-CHOP

Definition of primary breast DLBCL - Isolated breast involvement with or without nodal disease, which include distant nodal disease as well as regional nodal disease

Definition of nodal DLBCL

- The disease was only limited to the lymph nodes or lymphoid organs

Exclusion Criteria:

* Primary breast DLBCL or nodal DLBCL treated without rituximab
* Secondary breast DLBCL
* Recurrent DLBCL
* Stage III or IV of nodal DLBCL with extranodal involvement as a dissemination process

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary breast DLBCL group was identified from the nation-wide surveys in the university hospital, general hospital, and cancer institute of Korea. And, the nodal DLBCL group, as a matching control group, was selected from the data registry of Korean Society of Hematology Lymphoma Working Party.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 year

SECONDARY OUTCOMES:
Progression-free survival | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Kwak, MD.,PhD., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

REFERENCES:
- [Derived] Yhim HY, Kim JS, Kang HJ, Kim SJ, Kim WS, Choi CW, Eom HS, Kim JA, Lee JH, Won JH, Shim H, Huh J, Lee DH, Suh C, Kwak JY. Matched-pair analysis comparing the outcomes of primary breast and nodal diffuse large B-cell lymphoma in patients treated with rituximab plus chemotherapy. Int J Cancer. 2012 Jul 1;131(1):235-43. doi: 10.1002/ijc.26352. Epub 2011 Aug 30. PMID 21823120